CLINICAL TRIAL: NCT03164707
Title: Predictive ValueOf Admission Blood Glucose Level In Patients With ST-Segment Elevation Myocardial Infarction Undergoing Primary Percutaneous Angioplasty
Brief Title: Predictive Value Of Admission Blood Glucose Level In Patients With Acute Myocardial Infarction
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, George Motea Ghayes, Principal Investigator, Assiut University
Other Study IDs: Serum Blood Glucose Level
Record Dates: First submitted 2017-05-22; First posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Predictive Value of Admission Blood Glucose Level in Acute Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Blood Glucose Level — ON Admission Blood Glucose Level Fasting Blood Glucose Level

SUMMARY:
Coronary atherosclerosis is the leading cause of death worldwide. Diabetes mellitus is associated with increased prevalence of coronary artery disease

Increased plasma glucose is a common feature in the acute phase of myocardial infarction, even in patients without diabetes. Patients with stress hyperglycemia, but without previous diagnosis of diabetes, were at increased risk of congestive heart failure, arrhythmia and cardiogenic shock as well as increased both in-hospital and long-term mortality . Previous studies have demonstrated larger infarct size and poorer prognosis inpatients with hyperglycemia upon hospital admission compared with patients without hyperglycemia

It has been reported that stress hyperglycemia impairs microvascular circulation and may lead to no-reflow phenomenon. No reflow phenomenon was significantly more frequent among patients with hyperglycemia and increased progressively with increasing admission blood glucose in patients with Acute Myocardial Infarction . Furthermore, patients with high admission glucose are more likely to develop restenosis and require repeat revascularization procedures compared with those with normal admission glucose and are also at increased risk for repeated Myocardial Infarction, stent thrombosis and death.

ELIGIBILITY:
Inclusion Criteria:

acute ST Segment Elevation Myocardial Infarction patients not known to have Diabetes Mellitus undergoing primary PCI.

Exclusion Criteria:

* patients known to have Diabetes mellitus (known diabetes mellitus on admission, which was treated with diet, oral glucose-lowering medication, and/or insulin).
* Patients with prior Primary Percutaneous Intervention and/or Coronary Artery Bypass Graft (altering disease state).
* Patients with severe liver or renal disease (altering disease state).
* Patients with anemia, kidney disease or certain blood disorders (thalassemia).

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Acute ST Segment Elevation Myocardial Infarction admitted in Assiut University Hospital
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Correlation of level of blood glucose on admission in patients with ST Segment Elevation Myocardial Infarction and Hospital Outcome | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: George Motea Doos, M.B.B.CH, Principal Investigator — Assiut University

REFERENCES:
- [Result] Cura FA, L'Allier PL, Kapadia SR, Houghtaling PL, Dipaola LM, Ellis SG, Topol EJ, Brener SJ; GUSTO IIb and RAPPORT Investigators. Predictors and prognosis of suboptimal coronary blood flow after primary coronary angioplasty in patients with acute myocardial infarction. Am J Cardiol. 2001 Jul 15;88(2):124-8. doi: 10.1016/s0002-9149(01)01605-8. PMID 11448407
- [Result] Gearhart MM, Parbhoo SK. Hyperglycemia in the critically ill patient. AACN Clin Issues. 2006 Jan-Mar;17(1):50-5. doi: 10.1097/00044067-200601000-00007. PMID 16462409
- [Result] Iwakura K, Ito H, Ikushima M, Kawano S, Okamura A, Asano K, Kuroda T, Tanaka K, Masuyama T, Hori M, Fujii K. Association between hyperglycemia and the no-reflow phenomenon in patients with acute myocardial infarction. J Am Coll Cardiol. 2003 Jan 1;41(1):1-7. doi: 10.1016/s0735-1097(02)02626-8. PMID 12570936
- [Result] Mehta RH, Harjai KJ, Cox D, Stone GW, Brodie B, Boura J, O'Neill W, Grines CL; Primary Angioplasty in Myocardial Infarction (PAMI) Investigators. Clinical and angiographic correlates and outcomes of suboptimal coronary flow inpatients with acute myocardial infarction undergoing primary percutaneous coronary intervention. J Am Coll Cardiol. 2003 Nov 19;42(10):1739-46. doi: 10.1016/j.jacc.2003.07.012. PMID 14642681
- [Result] Rasoul S, Ottervanger JP, Bilo HJ, Timmer JR, van 't Hof AW, Dambrink JH, Dikkeschei LD, Hoorntje JC, de Boer MJ, Zijlstra F. Glucose dysregulation in nondiabetic patients with ST-elevation myocardial infarction: acute and chronic glucose dysregulation in STEMI. Neth J Med. 2007 Mar;65(3):95-100. PMID 17387235